CLINICAL TRIAL: NCT07183631
Title: Evaluating Treatment of Intra-bony Defects With PRF or EMD
Brief Title: Healing of Intrabony Defects Following Treatment With PRF or EMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Eleonora Solyom, Assistant Lecturer, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRF_EMD periodontal defect
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Periodontal Bone Loss; Periodontal Disease; Platelet Rich Fibrin
MeSH Terms: conditions — Alveolar Bone Loss; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet-rich fibrin (Experimental)
  Interventions: Other: Platelet rich fibrin
- Enamel matrix derivate (Sham Comparator)
  Interventions: Other: Enamel matrix derivate

INTERVENTIONS:
Other: Platelet rich fibrin — Platelet-rich fibrin (PRF) was prepared according to the manufacturer's instructions. A blood sample was collected from the cubital vein in 10 ml tubes without anticoagulant and centrifuged at 3000 rpm for 10 minutes using a GLO GT416 table centrifuge (GLO Glotech Co. Ltd, Korea) and GLO PRP collection kit (GLO PRP-Kit, Glotech Co, Asan Choong-nam, Korea/ Glofinn, Finland).
  Arms: Platelet-rich fibrin
Other: Enamel matrix derivate — In the control group, the root surface was conditioned with 24% ethylenediaminetetraacetic acid (EDTA) gel for two minutes, washed with physiological saline solution, dried, and treated with enamel matrix derivative (EMD), ("Emdogain", Straumann, Switzerland) per manufacturer recommendations.
  Arms: Enamel matrix derivate

SUMMARY:
Objective: To evaluate clinically the long-term results following treatment of deep intrabony defects with either platelet-rich fibrin gel (PRF) or an enamel matrix derivative (EMD).

Methods: Twenty six patients diagnosed with advanced chronic periodontitis, and each of whom displaying one deep intrabony defect were randomly treated with open flap debridement and with either PRF (test) or EMD (Emdogain, Straumann, Basel, Switzerland) (control). The clinical outcomes were evaluated at baseline, at six months and three years after treatment. The primary outcome variable was the clinical attachment level (CAL).

ELIGIBILITY:
Inclusion Criteria:

1. No systemic conditions affecting treatment outcomes
2. Good oral hygiene [plaque index (PI) <1; Löe 1967]
3. Compliance with the maintenance program
4. Presence of at least one intra-bony defect with a probing depth (PD) of ≥6 mm and an intra-bony component of ≥3 mm confirmed by radiographs.

Exclusion Criteria:

* significant medical conditions: irradiation in the maxillofacial area, uncontrolled diabetes or hypertension, systemic steroid or bisphosphonate treatment, pregnancy, or lactation, infectious diseases,
* age <18 years, (3) smokers (>5 cigarettes/day),
* high residual inflammation (FMBS >25%),
* poor oral hygiene (FMPS >25%), and
* defect-related factors: furcation involvement, endo-perio defects, horizontal defects, or multi-tooth defects .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth (PPD) | preop and after 6 months

SECONDARY OUTCOMES:
Gingival recession | preop and after 6 months
Clinical attachment loss | preop and after 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No